CLINICAL TRIAL: NCT05498974
Title: China Diabetes Type 1 Study (CD1S) by China Alliance for Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Director, National Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital of Central South University
Other Study IDs: CD1S
Record Dates: First submitted 2022-07-02; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Type1diabetes; Diabetes
Keywords: Type 1 diabetes; Diabetes in Young
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals diagnosed with type 1 diabetes: All patients diagnosed with type 1 diabetes of all ages.
  Interventions: Other: Standard type 1 diabetes management model constructed by China Alliance for Type 1 Diabetes in each center
- Individuals with diabetes who had an age of onset <= 20 years.: All patients with diabetes who had an age of onset <= 20 years.
  Interventions: Other: Standard type 1 diabetes management model constructed by China Alliance for Type 1 Diabetes in each center

INTERVENTIONS:
Other: Standard type 1 diabetes management model constructed by China Alliance for Type 1 Diabetes in each center — Standard type 1 diabetes management model constructed by China Alliance for Type 1 Diabetes in each center

SUMMARY:
The aim of the China Diabetes Type 1 Study (CD1S) is to conduct a nationwide type 1 diabetes (T1D) registry study in patients with T1D and in pediatric adolescent patients with diabetes who had an age of onset <= 20 years.

CD1S compromises a retrospective study enrolling inpatients hospitalized from Jan 1st, 2016 to Dec 31, 2021, and a prospective study beginning from the year 2022.

DETAILED DESCRIPTION:
The aim of the China Diabetes Type 1 Study (CD1S) is to conduct a nationwide type 1 diabetes (T1D) registry study to investigate the demographic characteristics, metabolic control, complications occurrence as well as risk factors of patients with T1D, and to investigate the clinical features, complications' burdens and risk factors in pediatric adolescent patients with diabetes who had an age of onset <= 20 years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with type 1 diabetes mellitus of any duration; meeting criteria (1) or any of (2) or any of (3)

  1. Clinical diagnosis of type 1 diabetes by a specialist
  2. Age at onset < 15 years; no overweight or obesity at onset; previous diabetic ketoacidosis; highest random C-peptide < 200 pmol/L
  3. Initiation and continuation of insulin therapy (except pancreatic or islet transplantation) after diagnosis; positive islet autoantibodies Or 2. Children and adolescents with diabetes mellitus at age of onset <= 20 years, regardless of type and duration of disease.

Exclusion Criteria:

* For enrolment of patients with T1D, exclusion was made if any of the following criteria were met (not applicable to those with onset under 20 years of age)

  * No insulin dependence for at least 6 months after diagnosis of diabetes mellitus.

    * No DKA for 1 month off insulin for those with a history of diabetes > 1 year. ③ C-peptide > 800 pmol/L at any time point.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 1 diabetes or children and adolescents with diabetes mellitus at age of onset <= 20 years
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum hemoglobin A1c level | Every year for up to 10 years
  A1c reflects the average blood glucose level
Albumin-to-creatinine ratio in urine sample | up to 10 years
  Albumin-to-creatinine ratio in urine sample
Arteriosclerotic cardiovascular diseases | up to 10 years
  Incident cases of cardiovascular diseases
Electromyography | up to 10 years
  value of nerve conduction velocity, F wave index, H-reflex
PHQ-9 | up to 10 years
  PHQ-9（a score between 0-27, ≥10 may indicate depression)
GAD-7 | up to 10 years
  GAD-7(a score between 0-21, ≥5 may indicate general anxiety)
WHO-5 | up to 10 years
  WHO-5 (a score between 0-100, higher score means better outcome)
PAID | up to 10 years
  PAID (a score between 0-100, ≥40 warrants special attention).

SECONDARY OUTCOMES:
Change in C-peptide | Every year for up to 10 years
  C-peptide are measured before and 2-hour after a mixed meal tolerance test at each follow-up of this study
Change in titer of autoantibodies | Every year for up to 10 years
  Glutamic acid decarboxylase antibody
Fasting blood glucose | Every year for up to 10 years
  the blood sugar level after fasting for eight hours
Systolic blood pressure | Every year for up to 10 years
  Systolic blood pressure
Diastolic blood pressure | Every year for up to 10 years
  Diastolic blood pressure
Change in lipid profiles | Every year for up to 10 years
  Including triglyceride, total cholesterol, HDL-cholesterol and LDL-cholesterol
Metabolomics | Every year for up to 10 years
  un-targeted metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, MD, PhD, Principal Investigator — The Second Xiangya Hospital, Central South University
Locations (11):
- China (11):
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - the First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Heji Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First People's Hospital of Yunnan, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No